CLINICAL TRIAL: NCT03829228
Title: An Evaluation of Proglucamune in the Treatment of Protective Qi
Brief Title: An Evaluation of Proglucamune in the Treatment of Protective Qi Insufficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USANA Health Sciences (Industry)
Collaborators: Elegant And Olive Health Clinic, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201875
Record Dates: First submitted 2018-12-18; First posted 2019-02-04 (Actual); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Protective Qi Insufficiency
Keywords: Protective Qi; Immunity

STUDY DESIGN:
Intervention Model Description: Subjects with Protective Qi Insufficiency
Masking Description: Given the small sample size in this pilot study and the potential drop-out rate, we did not include a placebo group to control for the placebo effect. Nonetheless, we implemented a "deceptive" double-blinding design, i.e., all on-site care-providers and investigators and all participants were told that this study was placebo controlled, and that each participant had a 50/50 chance of receiving treatment or placebo. This masking helps decreasing the expectation bias from the participants that confound the study result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proglucamune treatment (Experimental): Participants were treated with 2 tablets of Proglucamune per day for a total duration of 8 weeks.
  Interventions: Dietary Supplement: Proglucamune

INTERVENTIONS:
Dietary Supplement: Proglucamune — Following screening and enrollment, participants were treated with 2 tablets of Proglucamune per day for a total duration of 8 weeks. Each Proglucamune tablet contained ~100 mg ß-glucan derived from Baker's Yeast extract (Saccharomyces cerevisiae, cell wall), Reishi mushroom powder (Ganoderma lucidum), and Shitake mushroom powder (Lentinula edodes).

SUMMARY:
According to Traditional Chinese Medicine (TCM) principle, Protective Qi (PQi) is a one specific concept of Qi that provides the vital energy of the body. It works primarily on the body surface as a defensive barrier. In this context, PQi is analogous to anatomical barriers of the innate immune system located for example, at the skin surface and the mucosal surfaces of the respiratory and digestive tract. Individuals with PQi Insufficiency are predisposed to frequent cold and other symptoms caused by invasion of external pathogens ("Wai Xie" or "external evil" in TCM).

ß-glucan is a polysaccharide that activates macrophage (Dectin-1) and neutrophil (CR3) receptors, and therefore enhances immune defense at digestive and respiratory mucosa. Clinical trials have shown its immune activity such as preventing upper respiratory tract infection (URTI) and Traveler's diarrhea. Notably, ß-glucan is a component of Ganoderma Luciderm (or Reishi / Lingzhi), one TCM ingredient well-known for improving Qi. Based on this connection, investigators hypothesized that ß-glucan is the active ingredient in Reishi that at least partially accounts for Reishi's activity on Qi.

To test our hypothesis, investigators have conducted an uncontrolled pilot trial that investigated the effect of a commercially available, high ß-glucan containing product, Proglucamune®, on PQi status. Proglucamune contains ß-glucan from three different natural sources: Reishi mushroom, Shiitaki mushroom, and Bakers' yeast, each providing ß-glucan that differs slightly in their molecular structure. Through this pilot investigators sought to obtain an estimate of the effect size of Proglucamune on PQi that would allow us, via statistical methods, to estimate the necessary sample size for more definitive future trials.

DETAILED DESCRIPTION:
Unlike mainstream Western medicine (WM), alternative medicines (AM) such as Traditional Chinese Medicine (TCM), emphasizes individually-differentiated therapies. As such, AM therapies are normally not tested in clinical studies that statistically demonstrate the efficacy at the populational level for applicable patients, and this makes it difficult to objectively evaluate and compare different therapies. The lack of clinical studies stands as a barrier for the advance of AMs as well as their engagement with WM. In fact, most researchers view AMs primarily as untapped sources of "active ingredients/compounds" for drug development, but disregard the rationales under which the therapies were developed. A "One-Way-Traffic" research paradigm is thus created wherein AM therapies are investigated for their efficacy by WM standards, whereas the vast potential of employing WM therapies for AM therapeutics is ignored. In light of this, investigators set up a novel strategy that bridges TCM and WM, i.e., testing a WM-based therapy by TCM standards through clinical trial/statistics- based method.

Qi is a central concept of traditional Chinese medicine (TCM) and was first documented in the oldest TCM writings more than 2000 years ago. Generally speaking, Qi refers to the vital energy of the body and is derived from two primary sources: 1) inborn Qi (that may be construed as genetics), and 2) pectoral Qi (can be construed as metabolism). Moreover, Qi manifests itself in two forms: Nutritive Qi and Protective Qi, which can be understood to reflect an individual's nutritional state and immune health, respectively. Regarding the latter, protective Qi functions to defend the body from the invasion of external pathogens. TCM also emphasizes that Protective Qi works primarily on the body surface as a defensive barrier. In this context, Protective Qi is analogous to anatomical barriers of the innate immune system located for example, at the skin surface and the mucosal surfaces of the respiratory and digestive tract.

TCM has developed a number of methods to strengthen the Qi. Prominent among these is the use of Reishi, either alone or in combination with other TCM remedies. The use of Reishi was described in detail in the first TCM pharmacopeia "Compendium of Materia Medica" published in year 1,600. Nonetheless, although Protective Qi is part of the general Qi, the specific effect of Reishi on Protective Qi is less documented. Anecdotal reports are available that claim significant improvement of Protective Qi with Reishi or Reishi-containing formulas within days. Notably, Western medicine has identified immune-boosting properties of Reishi, which may explain the Qi enhancing effects of this plant. Specifically, beta-glucan - a component of Reishi - has been shown to activate macrophage (large white blood cells in the immune system that destroy bacteria and other harmful substances), neutrophil (type of white blood cells that are important for protection against infections), and other immunocytes (a type of cells capable of producing an immune response), and may exhibit particular benefits among macrophage-rich organs such as the lung, liver and spleen. In fact, ß-glucans from sources other than Reishi, such as baker's yeast, are able to initiate the same immune response and clinical benefits.

The overlap of TCM and western medicine concerning the beneficial effects of Reishi for its Qi enhancing and immune-modulating effects, respectively, has prompted us to investigate whether or not Reishi, in conjunction with other natural products used in TCM, can enhance an individual's Protective Qi. More specifically, the objective of the current protocol is to determine if a commercially available dietary supplement (Proglucamune®, USANA Health Sciences) containing powdered Reishi and Shitake mushrooms as well as baker's yeast extract, and which is comprised of 11% ß-glucans by weight, will improve Protective Qi in subjects diagnosed by practitioners of TCM as having low or insufficient Protective Qi. Specifically, in this a pilot study, investigators sought to obtain an estimate of the effect size of Proglucamune on PQi that would allow us, via statistical methods, to estimate the necessary sample size for more definitive future trials. The trial also aimed to provide information on individuals who are responsive to Proglucamune treatment (responder), and subsequently recruit targeted individuals for the follow-up trials.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females aged 18 to 65 years (inclusive) without regard to race or ethnic background
2. Provide a signed Informed Consent prior to entry in the study.
3. Willing to follow all study instructions and consume the assigned investigational product for 8 weeks.
4. Not currently taking a beta-glucan containing supplement or any other supplement that might interfere with the study design.
5. Ability to swallow tablets and pills.
6. Diagnosed as having Qi deficiency based on the following criteria:

   * exhibit a history of susceptibility to cold* (* as defined in Traditional Chinese Medicine, TCM)
   * exhibit a shortness of breath
   * exhibit a lack of energy or excessive fatigue
   * susceptible to spontaneous perspiration
   * exhibit a corpulent tongue with or without white fur
   * unwillingness to speak
   * weak or powerless pulse
   * pale complexion

Exclusion Criteria:

1. Persons diagnosed by TCM as having medical conditions other than low Qi.
2. Significant acute or chronic illness or other medical conditions that will prevent or interfere with giving an informed consent, or with participation in the study.
3. Persons with insulin-dependent and orally controlled diabetes will also be excluded from the study.
4. Scheduling difficulties or lack of transportation that will prevent or interfere with their ability to attend all of the necessary study visits.
5. Persons medically diagnosed with depression or anxiety disorders.
6. Persons with a history of alcohol abuse or other substance abuse within the previous 2 years.
7. Females who are attempting to become pregnant, pregnant, lactating or who have given birth within 1 year.
8. Persons who have had a medical surgery in the past 4 weeks.
9. Persons currently enrolled in a clinical trial, or who have completed a clinical trial within the last 4 weeks.
10. Allergies to mushrooms or other fungi.
11. Significant problems with constipation or diarrhea.
12. Persons exhibiting symptoms of cold* (*as defined by TCM) within the past 7 days.
13. A lifestyle or schedule incompatible with the study protocol.
14. Persons who are allergic to yeast products, have autoimmune disease/an immune disorder, or take antidepressants, blood thinners (anticoagulants), or immunosuppressant medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — participant eligibility is based on self-representation of gender identity.
Enrollment: 30 (Actual)
Dates: Start 2018-03-18 (Actual); Primary Completion 2018-06-03 (Actual); Study Completion 2018-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Bernstein, MD, Principal Investigator — Department of Family and Community Medicine, Humber River Hospital
Locations (1):
- Elegant And Olive Health Clinic, Markham, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan GC, Chan WK, Sze DM. The effects of beta-glucan on human immune and cancer cells. J Hematol Oncol. 2009 Jun 10;2:25. doi: 10.1186/1756-8722-2-25. PMID 19515245
- [Background] Bashir KMI, Choi JS. Clinical and Physiological Perspectives of beta-Glucans: The Past, Present, and Future. Int J Mol Sci. 2017 Sep 5;18(9):1906. doi: 10.3390/ijms18091906. PMID 28872611
- [Derived] Levy M, Wu JR, Shi JP, Cheng HJ, Qu XQ, Bernstein I, Sinnott R, Tian JQ. Proof-of-Concept and Feasibility Study to Evaluate the Effect of beta-Glucan on Protective Qi Deficiency in Adults. Chin J Integr Med. 2021 Sep;27(9):666-673. doi: 10.1007/s11655-020-3430-y. Epub 2020 Aug 19. PMID 32820452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the great Toronto area in Canada through advertisement and referral from other TCM practitioners. The enrollment was conducted at the Elegant and Olive Health Clinic at Markham, Canada. Subjects that met the criteria for inclusion were enrolled. The first participants was enrolled on March 18th,2018 and the last participant was enrolled in April 8th, 2018.
Pre-assignment Details: There was no wash-out or run-in period. All participants were assigned to received Proglucamune treatment. No participants were excluded before the start of treatment.
Groups:
- All Participants Received Proglucamune Treatment.: Following screening and enrollment, participants were treated with 2 tablets of Proglucamune per day for a total duration of 8 weeks. Each Proglucamune tablet contained ~100 mg ß-glucan derived from Baker's Yeast extract (Saccharomyces cerevisiae, cell wall), Reishi mushroom powder (Ganoderma lucidum), and Shitake mushroom powder (Lentinula edodes).
Period: Overall Study
Arm/Group | All Participants Received Proglucamune Treatment.
Started | 30
Completed | 29
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants were treated with 2 tablets of Proglucamune per day for a total duration of 8 weeks.
  Proglucamune: Following screening and enrollment, participants were treated with 2 tablets of Proglucamune per day for a total duration of 8 weeks. Each Proglucamune tablet contained ~100 mg ß-glucan derived from Baker's Yeast extract (Saccharomyces cerevisiae, cell wall), Reishi mushroom powder (Ganoderma lucidum), and Shitake mushroom powder (Lentinula edodes).
Arm/Group | All Participants
Number analyzed (Participants) | 29
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 47 [18 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 29
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 29
Medication [Count of Participants; unit: Participants]
  Yes | 5
  No | 24
Supplement [Count of Participants; unit: Participants]
  Yes | 10
  No | 19
Smoking [Count of Participants; unit: Participants]
  Yes | 0
  No | 29
Alcohol [Count of Participants; unit: Participants]
  Yes | 0
  No | 29

OUTCOME MEASURES:

1. Primary Outcome: Change of Protective Qi Score (PQS) Determined by a Standardized Assessment
Description: Protective Qi of each participant at baseline and each follow-up visit will be measured by an on-site investigator (licensed TCM practitioners) through a standardized quantitative assessment. The evaluation includes 3 health conditions relevant to PQD (cold frequency, symptoms, and signs). Each condition will be scored on a 1-10 scale based on a set of standardized criteria. The sub-scores will be weighted to arrive at a final PQS. So this PQS will be on a 1-10 scale, with 10 being the most healthy state. The change of the PQS from baseline, indicating the treatment effect, will be calculated and analyzed by statistical means.
Time Frame: The change of PQS was obtained by assessment of PQS at each follow-up visit from the baseline (start date). The follow-up visit was conducted every two weeks throughout the study, i.e., on the 14th, 28th, 42nd, and 56th day from the baseline.
Population: Intent to treat population(all participants assigned to treatment). Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 29
units on a scale
  Baseline | 6.3 (0.23)
  Visit2 | 6.8 (0.17)
  Visit3 | 7.17 (0.15)
  Visit4 | 7.27 (0.18)
  Visit5 | 7.64 (0.16)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, ANOVA — The threshold for statistical significance was p=0.01; Mean Difference (Net) = 1.31, 95% CI 2-sided [0.62 to 2.01] — Treatment Difference= Visit5-Baseline

2. Primary Outcome: Change of Protective Qi (PQi) Status Determined by Traditional TCM Assessment
Description: PQi of each participant at baseline and each follow-up visit was measured by on-site investigators (licensed TCM practitioners) through the traditional TCM assessment, which was diagnosed based on investigators' experience. The evaluation includes 3 health conditions relevant to Protective Qi Deficiency (cold history, symptoms, and signs) but was neither standardized nor quantitative. PQi status was characterized as non-PQD (i.e., healthy condition, no PQD detected) or PQD (i.e., unhealthy condition). The change of the PQi status from baseline, indicating the treatment effect, was analyzed by categorical statistic.
Time Frame: PQi status was determined at the baseline (start date) and each follow-up visit. The follow-up visit was conducted every two weeks throughout the study, i.e., on the 14th, 28th, 42nd, and 56th day from the baseline.
Population: Intent to treat population (all participants assigned to β-glucan treatment). Last observation carried forward (LOCF) imputation method.
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 29
Participants
  Baseline: Non-PQD | 9
  Baseline: PQD | 20
  Visit2: Non-PQD | 10
  Visit2: PQD | 19
  Visit3: Non-PQD | 11
  Visit3: PQD | 18
  Visit4: Non-PQD | 19
  Visit4: PQD | 10
  Visit5: Non-PQD | 27
  Visit5: PQD | 2
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, Regression, Logistic — The threshold for statistical significance was p=0.01

3. Secondary Outcome: Change of Generic Qi Score (GQS) Determined by a Standardized Assessment
Description: Generic Qi of each participant at baseline and each follow-up visit will be measured by an on-site investigator (licensed TCM practitioners) through a standardized quantitative assessment. The evaluation includes 5 sets of criteria indicative of Generic Qi insufficiency (cold history, symptoms of PQD, symptoms of Lung Qi Deficiency, symptoms of Heart and Spleen Deficiency, and signs of GQD). Each set will be scored on a 1-10 scales, with 10 being the most healthy state. The sub-scores will be averaged to arrive at a final GQS. So this GQS will be on a 1-10 scale, with 10 being the most healthy state. The change of the GQS from baseline, indicating the treatment effect, will be calculated and analyzed by statistical means.
Time Frame: The change of GQS was obtained by deduction of GQS at each follow-up visit from the baseline (start date). The follow-up visit was conducted every two weeks throughout the study, i.e., on the 14th, 28th, 42nd, and 56th day from the baseline.
Population: Intent to treat population (all participants assigned to β-glucan treatment. Last observation carried forward (LOCF) imputation method.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 29
units on a scale
  Baseline | 6.34 (0.21)
  Visit2 | 6.76 (0.16)
  Visit3 | 7.16 (0.14)
  Visit4 | 7.29 (0.17)
  Visit 5 | 7.65 (0.16)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, ANOVA — The threshold for statistical significance was p=0.01; Mean Difference (Net) = 1.31, 95% CI 2-sided [0.64 to 1.98] — Treatment difference=Visit5-Baseline

4. Secondary Outcome: Change of Generic Qi (GQi) Status Determined by Traditional TCM Assessment
Description: GQi of each participant at baseline and each follow-up visit was measured by on-site investigators (licensed TCM practitioners) through the traditional TCM assessment,which was diagnosed based on investigators' experience and expertise. The evaluation was made through cold history, symptoms and signs but was neither standardized nor quantitative. GQi was characterized as Generic Qi Deficiency (GQD; unhealthy state) or non-GQD (healthy state). The change of the GQi status from baseline, indicating the treatment effect, was analyzed by rank-based statistic.
Time Frame: GQi was determined at the baseline (start date) and each follow-up visit. The follow-up visit was conducted every two weeks throughout the study, i.e., on the 14th, 28th, 42nd, and 56th day from the baseline.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 29
Participants
  Baseline: Non-GQD | 4
  Baseline: GQD | 25
  Visit2: Non-GQD | 4
  Visit2: GQD | 25
  Visit3: Non-GQD | 8
  Visit3: GQD | 21
  Visit4: Non-GQD | 9
  Visit4: GQD | 20
  Visit5: Non-GQD | 19
  Visit5: GQD | 10
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < 0.0001, Regression, Logistic — The threshold for statistical significant was p=0.01

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Our treatment tablets are supplement. All participants don't have allege in rhinitis, pollinosis( hay fever), or asthma.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
Study limitations: First, this was not a randomized, placebo-controlled trial, so the observed effect size likely was inflated by uncontrolled confounders. Second, most participants were receptive to the healing effects of TCM, which may have lead to an overestimate of treatment effect. Lastly, the clinical trial started when flu season had passed its peak. This may have decreased the chance of subjects catching the flu and thereby have led to improved PQi independent of Proglucamune treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT03829228/Prot_SAP_000.pdf